CLINICAL TRIAL: NCT04667585
Title: Radiotherapy Dose De-escalation in HPV-Associated Cancers of the Oropharynx Using Metabolic Signature From Interim 18FDG-PET/CT
Brief Title: Radiotherapy Dose De-escalation in HPV-Associated Cancers of the Oropharynx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00105899
Record Dates: First submitted 2020-11-19; First posted 2020-12-14 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Oropharynx Cancer
Keywords: PET-CT
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants undergo either reduced radiation dose or standard radiation dose based on the metabolic signature from an Interim 18FDG-PET/CT
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Interim PET-CT with dose de-escalation (Experimental): Participants will receive an interim PET-CT approximately 2 weeks into radiation therapy.
  Interventions: Radiation: De-escalated radiation dose; Other: 18 fluorodeoxyglucose (FDG)-positron emission tomography (PET)-Computed Tomography (CT)
- Interim PET-CT with standard radiation (Active Comparator)
  Interventions: Radiation: Standard radiation dose; Other: 18 fluorodeoxyglucose (FDG)-positron emission tomography (PET)-Computed Tomography (CT)

INTERVENTIONS:
Radiation: De-escalated radiation dose — Reduced dose of radiation applied to remaining radiation therapy when favorable interim PET-CT signature is produced
  Arms: Interim PET-CT with dose de-escalation
Radiation: Standard radiation dose — Standard dose of radiation applied to remaining radiation therapy when favorable PET-CT signature is not produced
  Arms: Interim PET-CT with standard radiation
Other: 18 fluorodeoxyglucose (FDG)-positron emission tomography (PET)-Computed Tomography (CT) — The CT scan - also called computerized tomography or just CT - combines a series of X-ray views taken from many different angles to produce cross-sectional images of the bones and soft tissues inside the body. CT scans in planning radiation therapy are standard of care. A PET is a highly specialized imaging technique that uses short-lived radioactive substances (such as FDG a simple sugar labeled with a radioactive atom) to produce three-dimensional colored images of those substances functioning within the body. These images are called PET scans and the technique is termed PET scanning. PET scanning provides information about the body's chemistry not available through other procedures. Unlike CT or MRI (magnetic resonance imaging), techniques that look at anatomy or body form, PET studies metabolic activity or body function.
  Other Names: 18 FDG-PET/CT

SUMMARY:
The purpose of this study is to use intra-treatment 18FDG-PET/CT during definitive radiation therapy for human papillomavirus (HPV)-related oropharyngeal cancer (OPC) as an imaging biomarker to identify and select patients with a favorable response for chemoradiation dose de-escalation. This study will prospectively evaluate the clinical outcomes for patients undergoing dose de-escalation.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of squamous cell carcinoma of the oropharynx with p16-positive immunohistochemical staining and/or positive HPV in situ hybridization (ISH) and/or positive HPV PCR
* Stage I-III (AJCC 8th edition) with plan for concurrent chemotherapy per standard of care treatment
* Zubrod/ECOG score of 0-1
* Weight loss <10% in the 3 months prior to diagnosis
* ≥ 18 years of age
* No prior chemotherapy for their current cancer diagnosis

Exclusion Criteria:

* Prior radiotherapy to the head and neck
* Medical contraindications to radiation therapy
* Absence of gross disease on imaging prior to beginning radiation therapy
* Distant metastatic disease
* Medical contraindication to PET/CT
* History of active cancer other than non-melanoma skin cancer within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | from initiation of radiation therapy through study completion, an average of 2 years
  defined as the time between initiation of radiation treatment and the first documented recurrence of disease or death due to any cause as measured by medical record abstraction

SECONDARY OUTCOMES:
locoregional progression-free survival | from initiation of radiation therapy through study completion, an average of 2 years
  as measured by abstraction from the medical record
distant disease-free survival | from initiation of radiation therapy through study completion, an average of 2 years
  as measured by abstraction from the medical record
overall survival | from initiation of radiation therapy through study completion, an average of 2 years
  as measured by abstraction from the medical record
progression free survival correlation in PET/CT responders versus PET/CT non-responders | 2 years
  as measured by the difference in median Kaplan-Meyer values
Acute adverse events | 7 weeks
  as measured by the number of participants who experience dermatitis, mucositis, xerostomia, dysphagia, dysgeusia, neutropenia, thrombocytopenia, nausea, vomiting, renal toxicity, and hearing loss
Long term adverse events | 2 years
  as measured by the number of participants who experience xerostomia, dysphagia, dysgeusia, trismus, lymphedema, superficial soft tissue fibrosis, hypothyroidism and periodontal disease

CONTACTS AND LOCATIONS:
Overall Officials: Jared Robbins, MD, Principal Investigator — DUHS
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No